CLINICAL TRIAL: NCT06865885
Title: Study of Optimal LDL-C Value Enhancement With Inclisiran in Patients With Multiple Comorbidities in Which There Are Drug-Drug Interactions Limiting LDL-C Lowering
Brief Title: LDL-C Optimization Using Inclisiran in Patients in Which Drug-Drug Interactions Limit LDL Lowering
Acronym: SOLVE-LDL-C
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Pam Taub, MD, Professor of Medicine, Directior of Preventative Cardiology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 810920; 315668-00001 (Other Grant/Funding Number: Novartis, Investigator Initiated Study)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Drug Interactions; Primary Prevention; Cardiometabolic Syndrome; LDL-Cholersterol Lowering
Keywords: Statin intolerance; drug drug interaction; inclisiran; LDL-Cholesterol; polypharmacy; multiple comorbidities
MeSH Terms: conditions — Metabolic Syndrome | interventions — ALN-PCS

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to the inclisiran arm (n=50) or will continue with standard of care (n=50). The study will consist of 5 study visits (screening, baseline, 3 mo., 9 mo., and 12 mo.). Patients in the inclisiran arm will be treated with subcutaneous injection of inclisiran 284mg (baseline, 3 months, then 9 month visit) as add-on therapy to SOC lipid-lowering therapies. LDL-C (primary endpoint) along with other biomarkers will be measured at screening, baseline, 3 mo., 9 mo., and 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care, no intervention (No Intervention): Patients will continue the standard of care for lipid lowering as deemed appropriate by their medical team, no changes to lipid lowering therapy are permited during the study.
- Inclisiran Arm (Active Comparator): Patients in the intervention arm will be treated with a subcutaneous injection of inclisiran 284mg for three doses (baseline visit, 3 months, then 9 month visit) as add-on therapy to the standard of care for lipid lowering as determined by their medical team.
  Interventions: Drug: Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) in 1.5 mL

INTERVENTIONS:
Drug: Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) in 1.5 mL — The intervention arm will receive subcutaneous injection of inclisiran 284mg at the baseline visit, 3 months and 9 month visit.
  Arms: Inclisiran Arm

SUMMARY:
Drug-drug interactions often limit statin optimization in a population of patients prescribed cytochrome P3A4 inhibitors, which include immunosuppressive agents, protease inhibitors, and antifungals. These patients frequently have autoimmune conditions or rheumatologic disorders that require complex drug regimens and are often on low-dose statin therapy or no statin at all, resulting in suboptimal LDL levels despite increased cardiovascular (CV) risk.

There is an unmet clinical need to improve LDL levels in this vulnerable patient population, which faces increased CV risk due to underlying conditions that also contribute to polypharmacy and multiple drug-drug interactions. This study is a randomized, open-label trial evaluating subcutaneous inclisiran plus standard of care for LDL-C lowering in high-risk primary prevention patients with multiple comorbidities (e.g., Type II diabetes, liver disease, chronic kidney disease, autoimmune disease, solid-organ transplant) who are taking five or more medications in which drug-drug interactions prevent optimization of statin therapy.

DETAILED DESCRIPTION:
This is an investigator-initiated, single-site, open-label, randomized trial. The investigators will enroll up to 100 high-risk primary prevention patients with at least one comorbidity and an indication for additional lipid control (such as Type II diabetes with A1c ≤ 8.5%, subclinical atherosclerosis, or ASCVD risk of 7.5% or greater). Patients will be randomized 1:1 to the inclisiran arm (n ≥ 50) with standard of care or standard of care alone (n ≥ 50).

The study will consist of five study visits (screening, baseline, 3 months, 9 months, and 12 months). Patients in the inclisiran arm will receive a subcutaneous injection of inclisiran 284 mg for three doses (baseline, 3 months, and 9 months following randomization) as add-on therapy. LDL-C (the primary endpoint) along with other biomarkers will be measured at screening, baseline (inclisiran dose #1), 3 months (inclisiran dose #2), 9 months (inclisiran dose #3), and 12 months (labs only). Patients will also undergo medical history and medication review at each visit. Surveys will be completed at each visit during the study period.

Patients in the control arm (standard of care) will continue with their current lipid-lowering therapy. No adjustments will be made to lipid-lowering therapy during the course of the study. Participants will be aware of the group to which they have been randomized.

The primary objective is to determine the efficacy of inclisiran for LDL-C lowering in high-risk primary prevention patients with multiple comorbidities (e.g., Type II diabetes, autoimmune disease, liver disease, chronic kidney disease, solid-organ transplant) who are taking five or more medications in which drug-drug interactions prevent optimization of statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study, including potential randomization to injections.
* Age >18 and <85 years and able to provide self-consent.
* Taking five or more prescription drugs at the time of enrollment, of any type.
* Meets at least one of the following criteria:

  * Elevated 10-year ASCVD risk score ≥7.5% (based on the ACC/AHA ASCVD Risk Estimator Plus tool).
  * Evidence of subclinical atherosclerosis including:

Calcification in any vascular bed, including coronary arteries and aorta. Calcification of cardiac valves. Breast calcification. Carotid plaque that is not hemodynamically significant.

o Type II diabetes on a stable medical regimen with HbA1c <8.5%. Per American Diabetes Association guidelines, patients with Type II diabetes aged 40-75 years should be on a moderate-intensity statin.

Patients with documented partial or complete statin intolerance are eligible for enrollment.

* On maximally tolerated statin therapy (which can be no statin for patients with documented intolerance) and have suboptimal LDL levels:

  * For patients with Type II diabetes: LDL >70 mg/dL or non-HDL >120 mg/dL.
  * For other patients: LDL >90 mg/dL or non-HDL >120 mg/dL.
* Willing to adhere to the randomized study regimen, including subcutaneous injection of inclisiran.
* Agreement to adhere to lifestyle considerations (see Section 5.3) throughout the study duration.

Exclusion Criteria:

* Prior or current use of inclisiran.
* Known hypersensitivity or allergy to inclisiran or its components.
* Active liver disease or unexplained persistent elevations in liver enzymes (ALT or AST >3x upper limit of normal).
* History of rhabdomyolysis or severe muscle-related statin intolerance.
* Uncontrolled diabetes (HbA1c >8.5%).
* Active malignancy requiring systemic therapy.
* Recent major cardiovascular event (myocardial infarction, stroke, or hospitalization for unstable angina) within the past 3 months.
* History of organ transplant other than solid-organ transplant.
* Pregnancy or breastfeeding.
* Any condition that, in the opinion of the investigator, would make participation unsafe or interfere with study procedures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of LDL-Cholesterol | 12 months
  Percent Change in LDL-C from baseline to month 12 of treatment with inclisiran as add on to background lipid-lowering therapy that includes maximally tolerated statin.

SECONDARY OUTCOMES:
Change in Atherogenic Lipid Burden | 12 months
  Absolute and percent change in LDL particle number, apo B, non-HDL, and small dense LDL, lipoprotein(a), from baseline (Visit 1) to month 12 of treatment with inclisiran

OTHER OUTCOMES:
Patient-Reported Experience | 12 months
  Patient-reported outcomes and experiences determined by surveys at each visit (the Standardized Treatment Satisfaction Questionnaire with Medication Relationship of the total number of medications on adherence to lipid lowering therapy).
Incidence of Adverse Events | 12 months
  Incidence of adverse events occurring during treatment with inclisiran.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wilkinson, MD, Study Director — University of California, San Diego; Eric D Adler, MD, Study Chair — University of California, San Diego; Pam Taub, MD, Principal Investigator — University of California, San Diego; Antoinette Birs, MD, Study Director — University of California, San Diego
Locations (1):
- UC San Diego Altman Clinical and Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not expected to be shared due to privacy concerns, institutional policies, and regulatory considerations. However, the Principal Investigator may determine that certain de-identified data may be shared with other researchers on a case-by-case basis, subject to appropriate approvals and data use agreements.

REFERENCES:
- [Background] Wright RS, Ray KK, Raal FJ, Kallend DG, Jaros M, Koenig W, Leiter LA, Landmesser U, Schwartz GG, Friedman A, Wijngaard PLJ, Garcia Conde L, Kastelein JJP; ORION Phase III Investigators. Pooled Patient-Level Analysis of Inclisiran Trials in Patients With Familial Hypercholesterolemia or Atherosclerosis. J Am Coll Cardiol. 2021 Mar 9;77(9):1182-1193. doi: 10.1016/j.jacc.2020.12.058. PMID 33663735
- [Background] Budoff MJ, Kinninger A, Gransar H, Achenbach S, Al-Mallah M, Bax JJ, Berman DS, Cademartiri F, Callister TQ, Chang HJ, Chow BJW, Cury RC, Feuchtner G, Hadamitzky M, Hausleiter J, Kaufmann PA, Leipsic J, Lin FY, Kim YJ, Marques H, Pontone G, Rubinshtein R, Shaw LJ, Villines TC, Min JK; CONFIRM Investigators. When Does a Calcium Score Equate to Secondary Prevention?: Insights From the Multinational CONFIRM Registry. JACC Cardiovasc Imaging. 2023 Sep;16(9):1181-1189. doi: 10.1016/j.jcmg.2023.03.008. Epub 2023 May 24. PMID 37227328
- [Background] American Diabetes Association Professional Practice Committee. 10. Cardiovascular Disease and Risk Management: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S179-S218. doi: 10.2337/dc24-S010. PMID 38078592
- [Background] Iribarren C, Chandra M, Lee C, Sanchez G, Sam DL, Azamian FF, Cho HM, Ding H, Wong ND, Molloi S. Breast Arterial Calcification: a Novel Cardiovascular Risk Enhancer Among Postmenopausal Women. Circ Cardiovasc Imaging. 2022 Mar;15(3):e013526. doi: 10.1161/CIRCIMAGING.121.013526. Epub 2022 Mar 15. PMID 35290077
- [Background] Fox CS, Vasan RS, Parise H, Levy D, O'Donnell CJ, D'Agostino RB, Benjamin EJ; Framingham Heart Study. Mitral annular calcification predicts cardiovascular morbidity and mortality: the Framingham Heart Study. Circulation. 2003 Mar 25;107(11):1492-6. doi: 10.1161/01.cir.0000058168.26163.bc. PMID 12654605
- [Background] Otto CM, Lind BK, Kitzman DW, Gersh BJ, Siscovick DS. Association of aortic-valve sclerosis with cardiovascular mortality and morbidity in the elderly. N Engl J Med. 1999 Jul 15;341(3):142-7. doi: 10.1056/NEJM199907153410302. PMID 10403851
- [Background] Ray KK, Wright RS, Kallend D, Koenig W, Leiter LA, Raal FJ, Bisch JA, Richardson T, Jaros M, Wijngaard PLJ, Kastelein JJP; ORION-10 and ORION-11 Investigators. Two Phase 3 Trials of Inclisiran in Patients with Elevated LDL Cholesterol. N Engl J Med. 2020 Apr 16;382(16):1507-1519. doi: 10.1056/NEJMoa1912387. Epub 2020 Mar 18. PMID 32187462
- [Background] Raal FJ, Kallend D, Ray KK, Turner T, Koenig W, Wright RS, Wijngaard PLJ, Curcio D, Jaros MJ, Leiter LA, Kastelein JJP; ORION-9 Investigators. Inclisiran for the Treatment of Heterozygous Familial Hypercholesterolemia. N Engl J Med. 2020 Apr 16;382(16):1520-1530. doi: 10.1056/NEJMoa1913805. Epub 2020 Mar 18. PMID 32197277
- [Background] Wiggins BS, Saseen JJ, Page RL 2nd, Reed BN, Sneed K, Kostis JB, Lanfear D, Virani S, Morris PB; American Heart Association Clinical Pharmacology Committee of the Council on Clinical Cardiology; Council on Hypertension; Council on Quality of Care and Outcomes Research; and Council on Functional Genomics and Translational Biology. Recommendations for Management of Clinically Significant Drug-Drug Interactions With Statins and Select Agents Used in Patients With Cardiovascular Disease: A Scientific Statement From the American Heart Association. Circulation. 2016 Nov 22;134(21):e468-e495. doi: 10.1161/CIR.0000000000000456. Epub 2016 Oct 17. No abstract available. PMID 27754879
- [Background] Hughes JE, Waldron C, Bennett KE, Cahir C. Prevalence of Drug-Drug Interactions in Older Community-Dwelling Individuals: A Systematic Review and Meta-analysis. Drugs Aging. 2023 Feb;40(2):117-134. doi: 10.1007/s40266-022-01001-5. Epub 2023 Jan 24. PMID 36692678
- [Background] Moran CA, Collins LF, Beydoun N, Mehta PK, Fatade Y, Isiadinso I, Lewis TT, Weber B, Goldstein J, Ofotokun I, Quyyumi A, Choi MY, Titanji K, Lahiri CD. Cardiovascular Implications of Immune Disorders in Women. Circ Res. 2022 Feb 18;130(4):593-610. doi: 10.1161/CIRCRESAHA.121.319877. Epub 2022 Feb 17. PMID 35175848